CLINICAL TRIAL: NCT05361499
Title: A Controlled Human Pneumococcal Infection Model (PIM) Study
Acronym: PIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL79171.091.22
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-04

CONDITIONS: Streptococcus Pneumoniae Infection
Keywords: Controlled human infection model; Streptococcus pneumoniae; Asymptomatic infection; Colonization; Healthy adults
MeSH Terms: conditions — Pneumococcal Infections; Asymptomatic Infections | interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Single dose open label intervention study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Streptococcus pneumoniae 6B (Sp_6B) inoculated (Experimental)
  Interventions: Biological: Sp_6B; Drug: Amoxicillin 500 mg

INTERVENTIONS:
Biological: Sp_6B — Intranasal inoculation of Streptococcus pneumoniae serotype 6B, 160,000 colony forming units (CFU)
Drug: Amoxicillin 500 mg — Amoxicillin, 7 days, 2x 500 mg

SUMMARY:
Infection with Streptococcus pneumoniae (the pneumococcus) is the leading cause of pneumonia, bacterial meningitis and bacteraemia worldwide in the very young and the elderly. Although pneumococcal vaccines exist, they do not provide complete protection and new strategies to combat this pathogen are urgently needed. Asymptomatic infection of S. pneumoniae in the human nasopharynx precedes the development of pneumococcal disease. Previously, an Experimental Human Pneumococcal Carriage (EHPC) model has been developed at the Liverpool School of Tropical Medicine (LSTM). The current study entails to establish this model in healthy adults living in the Netherlands using the inoculation dose currently used at LSTM.

Healthy adult participants (M/F) will be inoculated intranasally with strain BHN418, a penicillin sensitive serotype 6B strain of S. pneumoniae that was previously isolated from a healthy carrier. Following inoculation, participants will be monitored and blood and nasal samples will be collected over a period of 28 ± 3 days. Participants will receive a course of amoxicillin to eradicate infection on or shortly after the last visit at day 28 ± 3, unless S. pneumoniae is not detected on both day 14 and 28 ± 3 post-inoculation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged ≥ 18 and < 50 years on the day of the baseline visit.
2. Participant is in good health as confirmed by review of medical history and physical examination.
3. Participant has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
4. Participant has a home address within the Netherlands.
5. Participant is fully conversant in the Dutch language
6. Participant is able to communicate easily by both mobile telephone and text messaging
7. Participant is available to attend all study visits.
8. Participant agrees to inform his/her general practitioner (GP), in case applicable, about participation in the study and signs a request to release any relevant medical information concerning possible contra-indications for participation in the study by the GP.
9. Participant agrees to provide access to information regarding the vaccination background
10. Participant agrees to provide a treating physician access to all study-related information and data in case an adverse event occurs
11. Participant is able to arrive within 3h at the Radboudumc at any time during the study participation and participant is able to arrive within 1h at the Radboudumc from his/her home address. The participant must have a home address and live in the Netherlands.
12. Participant is willing to take an antibiotic regiment after inoculation with S. pneumoniae according to the study protocol.
13. Participant has signed informed consent.
14. Participant is able to answer all questions of the pre-consent questionnaire correctly.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results.
2. Smoking: Any smoking event in the last month, including (e-)cigarette, joint, cigar and pipe
3. Previous pneumococcal vaccination or infection with the pneumococcus at screening or inclusion visit
4. Close physical contact with at risk individuals, i.e. children under 5 years of age, immunosuppressed adults, frail elderly, chronically ill individuals. Close physical contact is defined as:

   * living in the same household
   * having work-related contact
   * spending more than 1 hour/day together with an at risk individual at less than 1.5 meter distance.
5. Illness at screening visit, illness at baseline (including mild upper respiratory tract infection, common cold, running nose), acute illness within 3 days prior to inoculation
6. Any antibiotic treatment within 2 weeks before inoculation
7. For female participants: pregnancy, lactation or intention to become pregnant during the study. Female volunteers are required to use an effective form of contraception during this study.
8. Known hypersensitivity to or contra-indications (including co-medication) for use of penicillin
9. Receipt of any vaccinations in the two weeks prior to the start of the study (inoculation) or plans to receive any other vaccinations during the study period.
10. Participation in any other clinical study (unless observational) in the three months prior to the start of the study or during the study period.
11. Being an employee or student of the department of Laboratory Medicine, Radboudumc.
12. Any other condition or situation that would, in the opinion of the investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Percentage of volunteers infected with S. pneumoniae serotype 6B following inoculation. | up to 4 weeks after inoculation

SECONDARY OUTCOMES:
The number of participants with sollicited AEs that are related to infection | from the baseline visit (between day -1 and -6) till the end of the study (day 28 ± 3)
The number, type and severity of sollicited AEs that are related to infection | from the baseline visit (between day -1 and -6) till the end of the study (day 28 ± 3)
Number of sampling timepoints with S. pneumoniae culture-positive nasal wash samples post-inoculation | On day 3, 7, 14 and 28 after inoculation
Number of colony forming units (CFUs) per ml detected in nasal wash of infected participants at each sampling timepoint | On day 3, 7, 14 and 28 after inoculation
Concentrations of S. pneumoniae-specific antibodies in blood and mucosal samples at the various sampling time points | On day 3, 7, 14 and 28 after inoculation

OTHER OUTCOMES:
Bacterial load as determined by PCR of pneumococcal genes at each sampling time point | On day 3, 7, 14 and 28 after inoculation
Cellular responses in blood and mucosal samples at various timepoints | On day 3, 7, 14 and 28 after inoculation
Soluble mediators in mucosal or blood samples at various timepoints | On day 3, 7, 14 and 28 after inoculation
Expression level of host genes at various timepoints | On day 3, 7, 14 and 28 after inoculation
Expression level of S. pneumoniae genes at various timepoints | On day 3, 7, 14 and 28 after inoculation
Presence of species other than S. pneumoniae in nasal washes at various timepoints | On day 3, 7, 14 and 28 after inoculation

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided